CLINICAL TRIAL: NCT05144685
Title: A Randomized, Double Blind Controlled Study to Evaluate the Safety and Effectiveness of a Digital Therapeutic for Individuals With Suicidal Ideation and/or Suicide Attempts
Brief Title: A Study to Evaluate the Safety and Effectiveness of a Digital Therapeutic
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Data Safety Monitoring Board (DSMB) recommendation per Charter stopping rules. The study surpassed the pre-planned futility boundary.
Sponsor: Oui Therapeutics, Inc. (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-Oui-001; 2R42MH123357-02 (NIH)
Record Dates: First submitted 2021-11-11; First posted 2021-12-03 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Suicide, Attempted; Suicidal Ideation
MeSH Terms: conditions — Suicide, Attempted; Suicidal Ideation | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and research assessors will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Experimental App + Treatment as Usual (Experimental): This intervention will be for the treatment group
  Interventions: Device: OTX-202; Behavioral: Treatment as Usual
- Other App + Treatment as Usual (Experimental): This intervention will be for the control group
  Interventions: Device: OTX-000; Behavioral: Treatment as Usual

INTERVENTIONS:
Device: OTX-202 — Experimental Pscyhoeducation and Intervention App
  Arms: Experimental App + Treatment as Usual
Device: OTX-000 — Other Pscyhoeducation App
  Arms: Other App + Treatment as Usual
Behavioral: Treatment as Usual — Treatment as usual may include appointments with psychiatrists and other mental health clinicians, suicide risk assessment, supportive listening, crisis resources, clinician assessment, and referral to outpatient treatment.
  Other Names: TAU

SUMMARY:
The primary objective of this study is to assess the effectiveness of a digital intervention in reducing suicide attempts.

DETAILED DESCRIPTION:
This double blind, randomized controlled trial will evaluate effectiveness of two digital interventions among 391 participants. Study participation will start when participants sign consent. Participants and research assessors will be blinded to treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

1. Ages ≥18 years old
2. Patients recently hospitalized.
3. Owns a smartphone.
4. Willing and able to complete enrollment procedures.
5. Able to understand the nature of the study.
6. Able and willing to provide at least two verifiable contacts.

Exclusion Criteria:

1. Patients who have untreated psychosis or active psychosis
2. Patients who appear to be impaired by the use of alcohol or other substance(s)
3. Patients who sign, or have signed, an informed consent form to participate in any clinical research
4. Patients who upon clinical examination are cognitively impaired
5. Patients with a medical condition that may compromise, interfere, limit, effect or reduce the subject's ability to complete

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Columbia-Suicide Severity Rating Scale(C-SSRS) | Screening, Week 4, Week 8, Week 12, Week 24, Week 52, Week 78, Week 104
  The C-SSRS will be used to assess change in suicide behaviors at 8 separate time points from screening period to Week 104.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - UCDDenver / Denver Health, Denver, Colorado
  - Yale, New Haven, Connecticut
  - Common Spirit, Omaha, Nebraska
  - Northwell Health, Glen Oaks, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Harding Hospital, Columbus, Ohio

REFERENCES:
- [Derived] Bryan CJ, Simon P, Wilkinson ST, Allen MH, Perez J, Adler C, Moon K, Astorino L, Carpenter KM, Misquitta L, Brownlowe K, Khazem LR, Hay J, Starkey AG, Tartaglia J, Winston H, Simpson S, Dager AD, Feuerstein S. A Digital Therapeutic Intervention for Inpatients With Elevated Suicide Risk: A Randomized Clinical Trial. JAMA Netw Open. 2025 Aug 1;8(8):e2525809. doi: 10.1001/jamanetworkopen.2025.25809. PMID 40779267